CLINICAL TRIAL: NCT04463927
Title: The Effect of Non-nutritive Sucking on Pain During Examination for Retinopathy of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Tuba Koc Ozkan, Assistant Professor, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/2-16
Record Dates: First submitted 2020-07-01; First posted 2020-07-09 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The non-nutritive sucking is applied to the group during the examination for retinopathy of prematurity
  Interventions: Other: non-nutritive sucking
- Control Group (No Intervention): The non-nutritive sucking is not applied to the control group.

INTERVENTIONS:
Other: non-nutritive sucking — intervention group received a sterile gloved finger during the examination for retinopathy of prematurity
  Arms: Intervention Group

SUMMARY:
Aim: The aim of the study is to determine the effect of non-nutritive sucking on pain during examination for retinopathy of prematurity.

Method: The study is conducted as a randomized controlled trial. The population of the study is premature newborn who treatment in a neonatal intensive unit. The premature newborns divided into two groups as an intervention and control group according to randomization. After the randomization, non-nutritive sucking is applied to the intervention group. No method is applied to the control group.

DETAILED DESCRIPTION:
A topical anesthetic will be applied to all premature newborns 30 seconds before eye examination. Non-nutritive sucking is applied to the intervention group during the examination for retinopathy of prematurity. No method is applied to the control group during the examination for retinopathy of prematurity

ELIGIBILITY:
Inclusion Criteria:

* having an examination for retinopathy of prematurity for the first time,
* age was between 28-35 weeks

Exclusion Criteria:

- having no congenital anomalies

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile | 1 minute
  The primary outcome of the study is to evaluate the pain relief efficacy of non-nutritive sucking during examination for retinopathy of prematurity Premature Infant Pain Profile (PIPP).

CONTACTS AND LOCATIONS:
Overall Officials: Tuba KOÇ ÖZKAN, Principal Investigator — Adiyaman University
Locations (1):
- Adiyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No